CLINICAL TRIAL: NCT04603742
Title: Anakinra in Adults With Severe COVID-19 and Features of Cytokine Storm Syndrome: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Anakinra, COVID-19, Cytokine Storm
Acronym: SOBI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding did not go through
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-07022396
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Cytokine Storm; Mechanical Ventilation Complication
Keywords: Anakinra; Covid19; Mechanical Ventilation; Cytokine Storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study is a phase II double-blind, placebo-controlled, multicentered trial. Patients in the intervention arm will receive anakinra IV (N=85) 4 times a day for 7 days. The placebo arm will receive normal saline IV (N=85) 4 times a day for 7 days. The investigators will follow up with patients for up to 60 days.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anakinra IV (Experimental): Patients in the intervention arm will receive anakinra IV (N=85) 4 times a day for 7 days. The investigator will follow up with patients for up to 60 days.
  Interventions: Drug: Anakinra
- Normal Saline IV (Placebo Comparator): Patients in the placebo arm will receive normal saline IV (N=85) 4 times a day for 7 days. The investigator will follow up with patients for up to 60 days.
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Anakinra — 100 mg of Anakinra will be mixed with 100 mL of 0.9% saline solution for IV administration.
  Other Names: Anakinra IV
  Arms: Anakinra IV
Drug: 0.9% Saline — The placebo preparation will consist of a 100 mL of 0.9% saline solution without the addition of anakinra.
  Other Names: Saline IV
  Arms: Normal Saline IV

SUMMARY:
The clinical syndrome associated with infection of the Coronavirus Disease 2019 (COVID-19) is notable for its variable clinical expression. Infection and transmission of the virus by asymptomatic individuals have been noted and represent one end of the clinical spectrum, while multi-organ failure, particularly pulmonary failure, and death represent the most severe end of the clinical spectrum. In a recent study published from the investigator's institution about the first 393 patients with COVID-19, 77.1% had a fever, a mechanism driven by IL-1. This suggests that there may be an excess release of IL-1 present.

Cytokine storm syndrome (CSS) has been observed in patients with COVID-19 and has been proposed to contribute to the acute pulmonary failure that occurs. In distinct clinical settings, macrophage activation syndrome, elevated levels of pro-inflammatory cytokines, including IL-1, IL-6, and others, as well as elevations in laboratory indicators, including ferritin, CRP, d-dimer, and lymphopenia, have been observed. IL-1 production is induced in response to inflammatory stimuli and mediates various physiologic responses including inflammatory and immunological responses. Anakinra, a recombinant IL-1 receptor antagonist, has shown promise in treating CSS. It inhibits both IL-1-alpha and IL-1-beta. It is an FDA approved medication used in rheumatoid arthritis (RA) and Cryopyrin-Associated Periodic Syndromes (CAPS). Anakinra's ability to inhibit both IL-1 subtypes and short half-life makes it favorable to some experts. In the investigator's case-series, using anakinra in patients with COVID-19 showed promising in preventing the need for mechanical ventilation, and mortality subsequently.

This study will determine the efficacy of anakinra, an interleukin (IL) -1 receptor blocker, in reducing the need for mechanical ventilation and/or 28-day mortality among patients with COVID-19 who have features of CSS and severe respiratory failure. The investigators will test the hypothesis that the proportion of subjects with COVID-19, features of CSS, and severe respiratory failure (World Health Organization (WHO) category 4 or 5) alive and without having required mechanical ventilation at day 28 from randomization will be 18% higher among those that receive anakinra compared to those that receive a placebo. A secondary hypothesis is that the number of subjects alive at 60-days will be higher amongst those who receive anakinra compared to those who receive a placebo.

ELIGIBILITY:
Inclusion Criteria

1. An IRB approved written Informed Consent Form (ICF) is signed and dated by the subject or legal representative.
2. The subject or legal representative must be considered capable of understanding the study procedures to provide consent for participation according to the judgment of the Investigator.
3. Molecular diagnosis of SARS-CoV-2 infection within 14 days of screening assessment.
4. Radiographic evidence of pneumonia by either chest X-ray or computerized tomography (CT) scan of the chest if collected as part of the standard of care.
5. Age between 18-89 years of age at the screening visit.
6. The subject must fulfill the inclusion criteria for CSS:

   1. Fever documented ≥ 38 ˚C (from the time of admission to the hospital), or historical fever (patient-reported).

      AND
   2. Respiratory failure defined as:

   i.Requiring supplemental O2 of ≥ 4 L nasal cannula or more to maintain an O2 saturation ≥ 92%, within 36 hours of the requirement for that level of O2.24 (Individuals on continuous positive airway pressure (CPAP) or high flow nasal cannula will be allowed)

   AND

   c. Ferritin > 1000 ng/mL at the time of screening.
7. Not requiring mechanical ventilation or ECMO at Screening and Baseline Assessments.
8. ANC must be > 1 x 10^9/L before randomization
9. Platelet count must be ≥ 50 x 10^9/L before randomization.
10. Negative pregnancy test before randomization (women of childbearing age only).
11. GFR ≥ 30 mL/min based on the Modification of Diet in Renal Disease equation.
12. Subjects participating in studies for convalescent plasma or anticoagulation protocol for COVID-19 will be included as long as these are also open-label.

Exclusion Criteria

1. The subject is not expected to survive for more than 48 hours from screening, in the opinion of the investigator.
2. Subjects participating in studies for COVID-19 with immunomodulating drugs, will be excluded. See Section 4.3.1 for drugs or investigational drugs for COVID-19 not allowed in this study.
3. Subject is currently participating in another study with an investigational drug. Participation in observational studies is allowed.
4. Known hypersensitivity to anakinra or E. coli derived proteins.
5. Existence of other evidence that can explain pneumonia including but not limited to: Influenza A virus, Influenza B virus, bacterial pneumonia, fungal pneumonia, or mycobacterial infection.
6. Known or suspected active TB including those incompletely treated, or known latent TB not adequately treated.

   1. Known or suspected active TB including those incompletely treated.
   2. Exclude patients with known latent TB including those incompletely treated (patient reported).
7. Known human immunodeficiency virus (HIV) infection.
8. Culture confirmed active bacterial infection requiring antibiotic therapy.
9. Subjects who are: do not intubate (DNI) and/or do not resuscitate (DNR) will not be allowed in the study.
10. Subjects already on mechanical ventilation or on extracorporeal membrane oxygenation (ECMO).
11. Subjects with Eastern Co-operative Oncology Group (ECOG)/WHO system score ≥ 3 before their hospital admission.
12. Subjects with past or current lymphoproliferative disorder requiring current medical treatment (e.g., chemotherapy, radiotherapy) for these conditions.
13. Current or past history of a solid tumor including breast or prostate cancer requiring current medical treatment.
14. Subjects receiving other immunosuppressants.
15. Use of the following medications within 6 months of randomization:

    1. Tumor necrosis factor inhibitors
    2. Chronic IL-1 use such as canakinumab or anakinra.
    3. IL-6 inhibitors: Use of any IL-6
    4. Janus kinase inhibitors
    5. Bruton's tyrosine kinase inhibitor
    6. C-C Chemokine receptor type 5
    7. Disease-modifying anti-rheumatic drugs (DMARD), which include cyclosporine, tacrolimus, cyclophosphamide, mycophenolic acid, mycophenolate, penicillamine, azathioprine, methotrexate.
    8. Rituximab and abatacept

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects alive without having required mechanical ventilation | 28 days post randomization
  This will be measured among subjects with COVID-19, features of CSS, and severe respiratory failure (WHO category 4 or 5) who are alive and without having required mechanical ventilation 28 days post randomization.

SECONDARY OUTCOMES:
60-day mortality | 60 days post randomization
  Mortality of participants will be compared between those that received anakinra and those that did not.
Patient Hospitalization | 28 days post randomization
  The number of days of hospitalization in the anakinra group compared to placebo after randomization up to day 28.
Patient Mechanical Ventilation | 28 days post randomization
  The number of days with supplemental oxygen, with noninvasive ventilation or high-flow oxygen at day 28 after randomization in the anakinra group compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Y Navarro-Millan, MD, MSPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medcine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu L, Wang B, Yuan T, Chen X, Ao Y, Fitzpatrick T, Li P, Zhou Y, Lin YF, Duan Q, Luo G, Fan S, Lu Y, Feng A, Zhan Y, Liang B, Cai W, Zhang L, Du X, Li L, Shu Y, Zou H. Clinical characteristics of coronavirus disease 2019 (COVID-19) in China: A systematic review and meta-analysis. J Infect. 2020 Jun;80(6):656-665. doi: 10.1016/j.jinf.2020.03.041. Epub 2020 Apr 10. PMID 32283155
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Background] Dinarello CA. The history of fever, leukocytic pyrogen and interleukin-1. Temperature (Austin). 2015 Apr 14;2(1):8-16. doi: 10.1080/23328940.2015.1017086. eCollection 2015 Jan-Mar. PMID 27226996
- [Background] WHO. Coronavirus disease (COVID-19) Therapeutic Trial Synopsis. 2020; https://www.who.int/blueprint/priority-diseases/key-action/COVID19_Treatment_Trial_Design_Master_Protocol_synopsis_Final_18022020.pdf. Accessed May 8, 2020, 2020.
- [Background] Navarro-Millan I, Sattui SE, Lakhanpal A, Zisa D, Siegel CH, Crow MK. Use of Anakinra to Prevent Mechanical Ventilation in Severe COVID-19: A Case Series. Arthritis Rheumatol. 2020 Dec;72(12):1990-1997. doi: 10.1002/art.41422. Epub 2020 Nov 4. PMID 32602262